CLINICAL TRIAL: NCT00917397
Title: The Outcome of Treatment of Traumatised Refugees With Trauma-Focused Cognitive Behavioural Therapy and / or Antidepressants - a Randomised Controlled Trial
Brief Title: The Outcome of Treatment of Traumatised Refugees With Psychotherapy and/or Antidepressants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Caecilie Buhmann (Other)
Responsible Party: Sponsor-Investigator, Caecilie Buhmann, Dr, Psykiatrisk Center Gentofte
Organization: Psykiatrisk Center Gentofte (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTF1
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Traumatized refugee; treatment; antidepressants; psychotherapy; PTSD in traumatized refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- psychotherapy (Experimental): Trauma-focused cognitive behavioral therapy
  Interventions: Behavioral: trauma-focused cognitive behavioural therapy
- Drug (Experimental): drug treatment and psychoeducation
  Interventions: Drug: Sertraline
- Waiting list (No Intervention): subjects randomized to waiting list
- Combination (Experimental): Both drug and psychotherapy
  Interventions: Drug: Sertraline; Behavioral: trauma-focused cognitive behavioural therapy

INTERVENTIONS:
Drug: Sertraline — varies
  Arms: Combination; Drug
Behavioral: trauma-focused cognitive behavioural therapy — once a week
  Arms: Combination; psychotherapy

SUMMARY:
The purpose of the study is to investigate the effect of treatment of traumatized refugees with a diagnosis of Post-Traumatic Stress Disorder (PTSD). The existing evidence point towards antidepressants of the type SSRI and trauma-focused cognitive Behavioural Therapy being the most effective treatments of PTSD, but very little evidence of treatment effects exist for the group of multitraumatized refugees. This study therefore seeks to investigate the treatment effect of 6 months drug therapy with antidepressants (Sertraline and/ or Mianserine) and/or trauma-focused cognitive behavioral therapy. A total of 200 individual will undergo treatment. They will be randomized to 4 different groups: antidepressants, psychotherapy, a combination og drug and psychotherapy and a waiting list. Outcome measures include symptoms, life quality and function. Patients with a diagnosis of drug abuse or psychosis will not be included. The hypothesis is that a combination of antidepressants and psychotherapy will be more effective than either of the two treatment regimes on their own.

ELIGIBILITY:
Inclusion Criteria:

* Adult traumatised refugee with PTSD

Exclusion Criteria:

* psychosis and drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Score on Harvard Traume Questionnaire (PTSD) | before entry, after 6 months treatment and at follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatrisk Center Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Buhmann CB, Nordentoft M, Ekstroem M, Carlsson J, Mortensen EL. Long-term treatment effect of trauma-affected refugees with flexible cognitive behavioural therapy and antidepressants. Psychiatry Res. 2018 Jun;264:217-223. doi: 10.1016/j.psychres.2018.03.069. Epub 2018 Apr 4. PMID 29655114
- [Derived] Buhmann CB, Nordentoft M, Ekstroem M, Carlsson J, Mortensen EL. The effect of flexible cognitive-behavioural therapy and medical treatment, including antidepressants on post-traumatic stress disorder and depression in traumatised refugees: pragmatic randomised controlled clinical trial. Br J Psychiatry. 2016 Mar;208(3):252-9. doi: 10.1192/bjp.bp.114.150961. Epub 2015 Nov 5. PMID 26541687